CLINICAL TRIAL: NCT00277082
Title: Pharmacology Study of Aerosolized Liposomal 9-Nitro-20 (S)- Camptothecin (L9NC) in Patients With Metastatic or Recurrent Cancer of the Endometrium or the Lung (NSCLC)
Brief Title: Aerosolized Liposomal Camptothecin in Patients With Metastatic or Recurrent Cancer of the Endometrium or the Lung
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Claire Verschraegen, MD; Prinicpal Investigator, University of New Mexico - CRTC
Other Study IDs: 1302C
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2008-04

CONDITIONS: Corpus Uteri; Lung Cancer
Keywords: Metastatic or Recurrent Cancer of the Endometrium or the Lung (NSCLC); Aerosolized Liposomal 9-Nitro 20; Camptothecin (L9NC)
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — rubitecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, lung tissue, lung cancer tissue.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 9-NC in aerosol reservoir — Samples will be minced or centrifuged and L9NC extracted by chromatography. L9NC will be measured by HPLC or mass spectrometry
  Other Names: Liposomal-Nitro-20 (S)-Camptothecin

SUMMARY:
To determine the concentration of 9-nitrocamptothecin (9NC) in the alveolar fluid over time.

1.2. To determine the arterial concentration of 9NC administered by inhalation in comparison to venous and urine concentrations.

1.3. To determine the tumor concentration of 9NC administered by inhalation

DETAILED DESCRIPTION:
TREATMENT PLAN (25-28) Patients will be admitted to the GCRC for 25 hours.

Admission will be prior to the daily DLPC-9NC administration

Upon admission, patients will be asked to empty their bladder. Urine will be collected for 24 hours, and refrigerated. Upon completion of the collection, urine will be mixed, and a 20 ml aliquot frozen and preserved for further analysis.

A catheter will be placed in a peripheral vein, and in a peripheral artery, and appropriately heparinized.

Venous and arterial blood samples (7 ml per samples) will be drawn in heparinized green tops prior to DLPC-9NC administration, and at the following time points: 2, 5, 8, 12, and 24 hours. An additional 2 samples may be drawn at the PI discretion. (Total blood drawn: 84 ml + 14 ml)

During the GCRG hospitalization, a bronchoalveolar lavage (BAL) will be done according to standard practice once per patients. Patients will be divided in cohort of 6 (3 females and 3 males). Each cohort will undergo the BAL at a specific time point: within 30 minutes of the end of DLPC-9NC treatment, at 3 hours, 8 hours, and 24 hours.

In responding patients that may become surgical candidate for a curative resection, one DLPC-9NC treatment will be administered prior to surgery (within 5 hours). Surgery will proceed as per standard of care and patients will sign a regular surgical consent for surgical procedure. Along with the tumor removal, one sample of venous blood and of arterial blood will be drawn for comparison (total volume: 14 ml). Once the tumor specimen is removed, a piece will be kept in liquid nitrogen, along with a piece of normal lung tissue, for further analysis. Patients will need to sign the attached consent form to authorize the collection of specimens.

ELIGIBILITY:
For Endometrial:

Inclusion Criteria:

* All patients, 18 years of age or older, with metastatic and/or recurrent endometrial cancer or with mixed mesenchymal malignant tumors whose epithelial component is recurring, who have failed standard chemotherapy or hormonal regimens for their disease or who refuse recommended standard chemotherapy are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients much have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of >= 1,500 or cells/mm³ and platelet count > 100,000/mm³ and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine <= 1.5 x upper limit of normal.
* Patients must not have a known symptomatic respiratory disease other than cancer, and must have a pulmonary function test equal to >= 50% FEV1, >= 50% FEV1/FVC, >= 50% TLC, and >= 50% DLCO of predicted values.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Any criteria that is borderline and may lead to ineligibility will be reviewed by the PI, who may override the eligibility criteria, after receiving sponsor agreement, if entry into the study is deemed to potentially benefit the patient.

For Lung:

Inclusion Criteria:

* All patients, 18 years of age or older, with stage 3b, 4, or recurrent, nonresectable, non-small-cell lung carcinoma are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine <= 1.5 x upper limit of normal.
* Patients must not have a known symptomatic respiratory disease other than cancer, and must have a pulmonary function test equal to >= 50% FEV1, >= 50% FEV1/FVC, >= 50% TLC, and >= 50% DLCO of predicted values.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Any criteria that is borderline and may lead to ineligibility will be reviewed by the PI, who may override the eligibility criteria, after receiving sponsor agreement, if entry into the study is deemed to potentially benefit the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, 18 years of age or older, with metastatic and/or recurrent endometrial cancer or with mixed mesenchymal malignant tumors whose epithelial component is recurring, who have failed standard chemotherapy or hormonal regimens for their disease or who refuse recommended standard chemotherapy.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2003-08; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States